CLINICAL TRIAL: NCT02966067
Title: A Split Mouth, Randomised Controlled Trial to Compare the Efficacy of an Array of 2x3 Pyramidal Microneedles of 280µm Height Versus a Standard 30-gauge Dental Needle in the Delivery of Local Anaesthetic Solution for Dental Procedures
Brief Title: A Split Mouth Trial to Compare Microneedles vs. Standard Needles in Dental Anaesthetic Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: Tyndall National Institute (Unknown)
Responsible Party: Principal Investigator, Darius Sagheri, Director of Orthodontic Therapy, University of Dublin, Trinity College
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: DDUH2011/09/07
Record Dates: First submitted 2016-11-04; First posted 2016-11-17 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Dental Pain; Anesthesia, Local
Keywords: Microneedles; Dental Anaesthesia
MeSH Terms: conditions — Toothache

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microneedle Device (Experimental): Local Dental Anaesthetic Solution Delivery System: Microneedle device with an array of 2x3 pyramidal wet-etch silicone microneedles of 280µm height to inject anaesthetic solution.
  Interventions: Device: Microneedle Device (Experimental)
- 30-gauge Short Hypodermic Needle (Active Comparator): Local Dental Anaesthetic Solution Delivery System: Standard thirty-gauge short hypodermic needle to inject anaesthetic solution.
  Interventions: Device: 30-gauge Short Hypodermic Needle

INTERVENTIONS:
Device: Microneedle Device (Experimental) — Injection of 1.2ml of a standard local dental anaesthetic solution [1.2ml of 2% lidocaine and 1:80,000 epinephrine (lidocaine 20 mg/ml, epinephrine 12.5 mμ/ml)] at a rate of 1 mL/min.
  Other Names: Local Dental Anaesthetic Solution Delivery System
  Arms: Microneedle Device
Device: 30-gauge Short Hypodermic Needle — Injection of 1.2ml of a standard local dental anaesthetic solution [1.2ml of 2% lidocaine and 1:80,000 epinephrine (lidocaine 20 mg/ml, epinephrine 12.5 mμ/ml)] at a rate of 1 mL/min.
  Other Names: Local Dental Anaesthetic Solution Delivery System
  Arms: 30-gauge Short Hypodermic Needle

SUMMARY:
The study will be completed as a two part, prospective, single-centre, randomised controlled trial.

Five volunteers (dentists) will be recruited in the first part of the study to evaluate and examine the microneedle device and its use. Based on those qualitative findings (individual interviews and focus group) modifications to the microneedle device will be implemented before part two of the study commences.

Twenty volunteers will be enrolled in the second part of the study. A split mouth design will be used to compare the efficacy of an array of 2x3 pyramidal wet-etch silicone microneedles of 280µm height with a standard 30-gauge short hypodermic needle in the delivery of local dental anaesthetic solution. Quantitative and qualitative measurements of the pain experienced and the depth of anaesthesia achieved will be recorded and compared.

DETAILED DESCRIPTION:
The study will be completed as a two part, prospective, single-centre, randomised controlled trial.

Five volunteers (dentists) will be recruited in the first part of the study in order to evaluate and examine the microneedle device and its use. Based on those qualitative findings (individual interviews and focus group) modifications to the microneedle device will be implemented before part two of the study commences.

Twenty healthy male volunteers will be invited to participate in the second part of the study. Participants will be randomly assigned to receive a dental anaesthetic solution injection with a microneedle device (Group I) or with a standard thirty-gauge short hypodermic needles (Group II) in the first week of the second part of the study.

Group I: The microneedle device will be applied randomly to the left or right buccal mucosa of the ﬁrst premolar tooth in the maxilla in order to inject slowly a standard local dental anaesthetic solution.

Group II: A standard thirty-gauge short hypodermic needles will be used for insertion and injection of the same standard local dental anaesthetic solution randomly to the left or right buccal mucosa of the ﬁrst premolar tooth in the maxilla.

Quantitative and qualitative measurements of the pain experienced and the depth of anaesthesia achieved will be recorded for both groups and compared.

In order to eliminate any carryover effects, a washout period of one week between receiving a second, opposite injection will be applied (i.e. Group I will receive an injection with a standard thirty-gauge short hypodermic needles and Group II an injection with the microneedle device). The buccal mucosa of the ﬁrst premolar tooth in the untreated, opposite maxilla side will receive an injection with the remaining injection method following the same procedure as described for the first week.

ELIGIBILITY:
Inclusion Criteria:

•Individuals are considered eligible for the study if they are not taking any medications and are deemed competent to complete the McGill pain questionnaire short-form (MPQ-SF) and visual analogue scale (VAS).

Exclusion Criteria:

* Individuals will be excluded from the study if they suffer from the following conditions:

  * Hypersensitivity to anaesthetics of the amide type
  * Epilepsy
  * Hypertension, impaired cardiac conduction
  * Impaired respiratory function
  * Impaired hepatic function
  * Cerebrovascular insufficiency
  * Thyrotoxicosis
* Interventions not permitted during the study include the use of steroids, analgesics or other non-steroidal inflammatory drugs and smoking.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-08 (Actual)

PRIMARY OUTCOMES:
Pain Evaluation | Immediately after injection of the anaesthetic
  Discomfort / pain intensity rating will be recorded by using a visual analogue scale (VAS)

SECONDARY OUTCOMES:
Pain Experience | Immediately after injection of the anaesthetic
  Discomfort / pain experience will be recorded by using the Short-Form McGill Pain Questionnaire
Electronic Pulp Test | 15 minutes after injection
  An electric pulp tester will be used to determine onset and duration of pulpal anaesthesia
Thermal Pulp Test | 10 minutes after injection
  Dental refrigerant spray will be sprayed on a cotton pellet and then applied to determine onset and duration of pulpal anaesthesia
Pin-Prick Test | 2 minute intervals alternating with fine touch test until onset of soft tissue anaesthesia
  Sensitivity of the buccal mucosa will be assessed with a spring algesimeter
Fine Touch Test | 2 minute intervals alternating with pin-prick test until onset of soft tissue anaesthesia
  Von Frey hair fibres will be used to evaluate the soft tissue sensitivity to touch

CONTACTS AND LOCATIONS:
Overall Officials: Darius Sagheri, Principal Investigator — University of Dublin, Trinity College; Ciarán P Devine, Principal Investigator — University of Dublin, Trinity College; June H Nunn, Principal Investigator — University of Dublin, Trinity College; Erica Donnelly-Swift, Principal Investigator — University of Dublin, Trinity College
Locations (1):
- University of Dublin, Trinity College, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No